CLINICAL TRIAL: NCT06142942
Title: Effect of Sprint Interval Training Frequency on Cardiorespiratory Fitness Adaptations
Brief Title: Effect of Sprint Interval Training Frequency on Improvements in Fitness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Tom Hazell, Principal Investigator, Wilfrid Laurier University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMRL-23-01
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Cardiorespiratory Fitness
Keywords: sprint interval training; maximal oxygen consumption; training intervention

STUDY DESIGN:
Intervention Model Description: Following pre-testing participants are assigned to one of the four groups based on their baseline cardiorespiratory fitness to ensure no differences between groups at baseline. Participants will train 2, 3, or 4 days a week, or be assigned to the control group (no training) and re-test following the 4 week intervention.
Who Masked: Outcomes Assessor
Masking Description: All pre- and post-testing is completed by researchers not involved in training, and thus are blinded to which group participants are assigned to. This prevents any potential bias when researchers are completing post-testing sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2 days per week group (Experimental): Participants in this group complete 2 training sessions each week (Monday and Thursday).
  Interventions: Other: Exercise Intervention
- 3 days per week group (Experimental): Participants in this group complete 3 training sessions each week (Monday, Wednesday, and Friday).
  Interventions: Other: Exercise Intervention
- 4 days per week group (Experimental): Participants in this group complete 4 training sessions each week (Monday, Tuesday, Thursday, and Friday).
  Interventions: Other: Exercise Intervention
- No-exercise Control group (No Intervention): This group does not complete any training intervention. They are asked to maintain their regular physical activity habits.

INTERVENTIONS:
Other: Exercise Intervention — Participants will complete an exercise intervention where they will exercise 2, 3, or 4 days per week for 4 weeks.
  Arms: 2 days per week group; 3 days per week group; 4 days per week group

SUMMARY:
The goal of this study is to learn how the number of weekly exercise sessions affects improvements in fitness in healthy university aged students. The main question it aims to answer is how training frequency affects improvements in fitness. Participants will complete a pre-testing sessions to assess fitness level and sprint performance. Following this participants are assigned to one of four groups. A group that exercises 2 days a week, a group that trains 3 days a week, a group that trains 4 days a week, or a no-exercise control group. Participants in this group will not complete any training and allow the researchers to compare the exercise groups to a group that didn't train. Each participant will train for 4 weeks. During each training session participants will complete 4-6 30 second all-out sprints with 4 minutes of rest between each. Participants will complete the same tests they did during the pre-testing session following the 4 weeks of training to see how frequency affects improvements.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active: exercising at least 2-3 days per week and not currently involved in, or had been involved in a systematic training program for at least 3 months prior to data collection.
* Safe to become physically active based on the Canadian Society for Exercise Physiology - Get Active Questionnaire.

Exclusion Criteria:

* Smoking
* Consuming supplements known to affect metabolism (e.g., creatine, carnitine, nitric oxide, brain chain amino acids).
* Failure to meet inclusion criteria

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | This will be assessed before and after 4 weeks of training (or control).
  Cardiorespiratory fitness will be assessed through the measurement of maximal oxygen consumption. This will be determined using an incremental exercise test to volitional fatigue on a treadmill. A metabolic cart will be used to assess oxygen consumption using indirect calorimetry

SECONDARY OUTCOMES:
Anaerobic performance | This will be assessed before and after 4 weeks of training (or control).
  Anaerobic performance will be assessed during one 30 second "all-out" sprint completed on a self-propelled treadmill. Participants will be instructed to run as fast and as hard as they can for the entire 30 seconds. Speed will be recorded during this sprint and used to determine, peak, average, and minimum speed, as well as fatigue index.

CONTACTS AND LOCATIONS:
Overall Officials: Tom J Hazell, PhD, Principal Investigator — Wilfrid Laurier University
Locations (1):
- Wilfrid Laurier University, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available to other researchers upon reasonable request.